CLINICAL TRIAL: NCT05053282
Title: Active Aging: Effect of Life-long Endurance Exercises on the Circadian Regulation of Physiological Processes and Their Maintenance in Aging
Brief Title: Long-life Endurance Exercise and Healthy Aging
Acronym: CAA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Comenius University (Other)
Collaborators: Physiko- und Rheumatherapie Gesellschaft m.b.H. (Unknown); University of Padova (Other); University of Roma La Sapienza (Other); University of Primorska (Other)
Responsible Party: Sponsor
Other Study IDs: 305041X157
Record Dates: First submitted 2021-08-03; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Aging
Keywords: aging; exercise; endurance running; circadian; inflammation; bone density
MeSH Terms: conditions — Motor Activity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood white cells blood serum and plasma skeletal muscle tissue from m. vastus medialis saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- master endurance athletes: men aged 65 to 75 with more than 150 minutes of running activity per week at least 15 years history of running
  Interventions: Other: endurance running exercise
- elderly sedentary: men aged 65 to 75 with no history of regular physical activity training and no more practice than 150 minutes of moderate or 75 minutes of vigorous intensity per week according the ACSM recommendations
- young endurance athletes: men aged 20 to 30 with more than 150 minutes of running activity per week at least 3 years history of running
  Interventions: Other: endurance running exercise
- young sedentary: men aged 20 to 30 with no history of regular physical activity training and no more practice than 150 minutes of moderate or 75 minutes of vigorous intensity per week according the ACSM recommendations

INTERVENTIONS:
Other: endurance running exercise — regular competitive or non-competitive running of medium and/or high intensity with the duration at least 20 minutes per session
  Groups: master endurance athletes; young endurance athletes

SUMMARY:
The project aims to explore the mechanisms by which lifelong exercise can promote healthy aging and slow down the negative impact of aging on the muscular system, immunity and the circadian system. The main goal of the project is to investigate the effect of lifelong endurance exercise on physical fitness, body composition, bone density and selected hormonal, biochemical, histological and molecular indicators of metabolic health and circadian clock function based on blood, immune cell and skeletal muscle tissue analyses in volunteers differentiated by age and weekly volume of physical activity.

It is hypothesized that lifelong endurance exercise may have beneficial effects on the circadian system stability and many, but not all health outcomes. Osteopenia/osteoporosis and low-grade malnutrition may be more prevalent in the group of endurance-trained senior runners.

In order to achieve the above research aims, sixty male subjects in total will be recruited according to inclusion and exclusion criteria. Four groups of subjects will differ according to their age and physical activity levels:

* a group of endurance-trained seniors (age range 65 - 75 year old, n=15) ● a group of sedentary seniors (age range 65 - 75 year old, n=15)
* a group of well endurance-trained young men (age range 20 - 30 year old, n=15) ● a group of sedentary young men (age range 20 - 30 year old, n=15).

Subjects must meet the following inclusion criteria:

1. for athletes' groups: defined as more than 150 minutes of running activity per week; for young athletes at least 3 years and for master athletes at least 15 years history of running.
2. for groups less active than recommended: no history of regular physical activity training and no more practice than 150 minutes of moderate or 75 minutes of vigorous intensity per week.

The standard inclusion criterion for every group will be body mass index (range 18.5-30 kg/m2).

No experimental study has been published on the potential of life-long exercise to attenuate the aging-induced disorganization of the circadian system and thus to promote healthy aging. In this aspect, the proposed study is original and up-to-date. Moreover, also other aspects of the study, e.g. exercise and inflammaging or the risks (besides the benefits) of the long-life endurance training on bone tissue etc. have been studied only scarcely. Therefore, more scientific information is needed before it can be safely prescribed to the aging population

ELIGIBILITY:
Inclusion Criteria:

for athletes' groups (master - 65 - 75 years old, and young athletes - 20 - 30 years old)

* more than 150 minutes of running activity which is by ACSM considered as vigorous intensity of endurance running for young athletes at least 3 years and for master athletes at least 15 years
* body mass index (BMI index) - range 18.5-30 kg/m2

for groups less active than recommended (sedentary young and elderly)

* no history of regular physical activity training and no more practice than 150 minutes of moderate or 75 minutes of vigorous intensity per week
* body mass index (BMI index) - range 18.5-30 kg/m2

Exclusion Criteria

* recent or current infection
* malignant disease
* uncontrolled hypertension (higher than 160 / 95mmHG)
* congestive heart failure (NYHA grade III and IV)
* unstable angina pectoris
* recent myocardial infarction (during the last 6 months)
* severe cardiac arrhythmia (anamnestic)
* chronic obstructive pulmonary disease
* presence of severe pulmonary, pleural or pericardial disease
* severe asthma
* recent sudden stroke (during the last 6 months)
* epilepsy
* insulin-dependent diabetes mellitus
* unstable bone lesions with a high risk of fractures
* other chronic diseases, at the discretion of the responsible doctor
* states of mental incompetence (severe anxiety and depression, dementia, alcoholism , or other dependencies, mental retardation)
* conditions complicating regular physical activity (uncontrollable pain, severe arthritis, planned knee / hip endoprosthesis, pathological fractures (last 6 months), amputation, use of walker, wheelchair
* pharmacological interference (e.g., steroids, nonsteroidal anti-inflammatory agents, immunosuppressive and antineoplastic drugs, beta blockers, statins)
* the use of performance-enhancing drugs in the past and during the study period

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inhabitants of Bratislava city (Slovakia) and those living within one hour drive by car from the laboratory (Faculty of Physical Education and Sport, Comenius University in Bratislava)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
maximal oxygen consumption | cross-sectional, one-point assessment over 1 day
  peak oxygen consumption normalised to body mass (mL/kg/min), measured through a graded cycling ergometry

SECONDARY OUTCOMES:
body composition | cross-sectional, one-point assessment over 1 day
  DXA method - fat mass (grams), lean mass (grams) and total mass (grams)
bone mineral content | cross-sectional, one-point assessment over 1 day
  DXA method - BMC (grams)
bone mineral density | cross-sectional, one-point assessment over 1 day
  DXA method - BMD (g/cm2)
maximum isometric muscle strength | cross-sectional, one-point assessment over 1 day
  maximum voluntary contraction (Nm) of both isometric extension and flexion on knee dynamometer
maximum isometric muscle torque development | cross-sectional, one-point assessment over 1 day
  rate of torque development (Nm/s) of both isometric extension and flexion on knee dynamometer
Immunohistochemical analyses - skeletal muscle cell morphometry | cross-sectional, one-point assessment over 1 day
  cross-sectional area (um2) of myosin heavy chain I (BA-D5) positive fibers
Immunohistochemical analyses - skeletal muscle tissue morphology | cross-sectional, one-point assessment over 1 day
  number of myonuclei, satellite cells, capillaries - counted per each fiber type nuclear number per fiber
circadian system phase | cross-sectional, two-point assessment at morning and afternoon over 1 day
  CD14-positive monocytes (mRNA levels of selected clock and clock-controlled genes /alternatively microarray analysis in sub-sample of subjects from each group) blood count

OTHER OUTCOMES:
skeletal muscle tissue - (PCR) RNA expression | cross-sectional, one-point assessment over 1 day
  Target genes for inflammatory markers
biochemical biomarkers of nitrogen compounds | cross-sectional, one-point assessment over 1 day
  creatinine (umol/L), total bilirubin (umol/L),uric acid(umol/L)
biochemical biomarkers of lipid and carbohydrate metabolism | cross-sectional, one-point assessment over 1 day
  serum glucose (mmol/L), total cholesterol urea (mmol/L), low-density lipoprotein cholesterol urea (mmol/L), high-density lipoprotein cholesterol urea (mmol/L), triacylglycerols (mmol/L)
biochemical malnutrition biomarkers | cross-sectional, one-point assessment over 1 day
  transthyretin, retinol binding protein(μg/mL)
biochemical liver function biomarkers | cross-sectional, one-point assessment over 1 day
  aspartate aminotransferase (ukat/L), alanine aminotransferase (ukat/L), γ-glutamyltransferase (ukat/L)
dietary macronutirents intake tracking | cross-sectional, one-point assessment over seven consecutive days
  Macronutrients (carbohydrate, fat, and protein in grams) data will be retrieved from each participant's diary and expressed as a daily average for total intakes.
dietary energy intake tracking | cross-sectional, one-point assessment over seven consecutive days
  Energy (kilocalorie) data will be retrieved from each participant's diary and expressed as a daily average for total and relative intakes.
physical activity monitoring | cross-sectional, one-point assessment over seven consecutive days
  ActivPAL device - static and dynamic acceleration to distinguish body posture as sitting/lying, standing, and stepping and estimate energy expenditure expressed as metabolic equivalents - MET
chronotype | cross-sectional, one-point assessment over 1 day
  score in The Munich ChronoType Questionnaire (MCTQ), total scores can range from 16 to 86, with the lowest values representing extreme-late chronotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Ján Cvečka, PhD., Principal Investigator — Comenius University
Locations (1):
- Comenius University in Bratislava, Faculty of physical education and sport Bratislava, Slovakia, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No